CLINICAL TRIAL: NCT03376243
Title: A Pilot Study to Determine the Feasibility of Early Emollient Use in Children With High Risk for Atopic Eczema - EARLYemollient
Brief Title: EARLYEMOLLIENT - Feasibility of Early Emollient Use in Children With Atopic Eczema
Acronym: EARLYemo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Prof. Dr. Stephan Weidinger, Deputy Head, Department of Dermatology and Allergy, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Earlyemollient Version 2.0
Record Dates: First submitted 2017-12-06; First posted 2017-12-18 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic eczema, prevention
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emollient (LIPIKAR BAUME AP+) (Experimental): Daily application of Lipikar Baume AP+ emollient AND Structured parent education
  Interventions: Other: LIPIKAR BAUME AP+ emollient
- Control (No Intervention): Only structured parent education

INTERVENTIONS:
Other: LIPIKAR BAUME AP+ emollient — Structured education on prevention guidelines
  Arms: Emollient (LIPIKAR BAUME AP+)

SUMMARY:
The aim of this pragmatic, parallel group, assessor-blind randomised open-label prospective study is to determine the reasons that motivate parents to enrol or not enrol their child in a randomized, controlled basic emollient trial for the prevention of atopic eczema (AE). Furthermore, this trial intends to test the hypothesis that daily skin barrier enhancement with Lipikar Baume AP+® in newborns at high risk is safe and efficient in preventing AE.

T

DETAILED DESCRIPTION:
The aim of this trial is to determine the reasons that motivate parents to enrol or not enrol their child in a randomized, controlled basic emollient trial for the prevention of AE. Furthermore, this trial intends to test the hypothesis that daily skin barrier enhancement with Lipikar Baume AP+® in babies at high risk of allergic disease is safe and to estimate the preventive effectiveness of Lipikar Baume AP+® in the prevention of AE in a high risk population.

Objectives:

The primary objectives are to investigate the

1. Feasibility:

   1. Parental willingness to enter a child in a controlled primary prevention trial
   2. Compliance with intervention
2. Safety: incidence of skin-related adverse events and serious adverse events during the study
3. Effectiveness:

   1. Cumulative incidence of AE within 2 years after randomization.
   2. Age of onset of AE

Study design:

Pragmatic, parallel group, assessor-blind randomised open-label prospective study of emollient use in 50 high-risk neonates starting between days 1 and 21. Child participation in the main part of the trial will be 2 years (from within 3 weeks of birth until approximately the child's second birthday). This will comprise a 1 year intervention phase then the primary outcome is assessed at 2 years.

Participants:

Participants will be newborn babies at high risk of developing AE defined as a parent or sibling who has (or had) doctor diagnosed asthma, AE or allergic rhinitis.

Intervention:

The intervention is daily application of emollient to the baby's entire body surface area including the face for the first year of life. Intervention and control group will receive structured parent education that comprises general advice on best practice skin care for their baby in line with the German AWMF S3 guidelines for allergy prevention and the Federal Centre for Health Education.

Data collection:

Infants will be examined at scheduled visits at Months 1, 6, 12, and 24. Telephone visits were performed at months 3 and 18 to assess for side effects, rashes, and compliance. Daily parental recordings will be assessed using electronic data capturing tools.

Primary Outcomes:

The primary outcomes will be feasibility, safety and tolerability, and preventive effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Participant (i.e. the newborn baby) must have a parent or sibling with a history of AE, allergic rhinitis or asthma.
* Infant in overall good health.
* Term-born babies
* Mother at least 18 years of age at delivery and capable of giving informed consent.

Exclusion Criteria:

* Preterm birth (defined as birth prior to 37 weeks gestation).
* Previous child randomised to this trial.
* Major congenital anomaly.
* Significant inflammatory skin disease at birth (except seborrheic dermatitis).
* Any immunodeficiency disorder or severe genetic skin disorder.
* Any condition that would make the use of emollients inadvisable or not possible.

Ages: 1 Day to 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Willingness to participate | 2 years
  Willingness of parents to get their child randomized and to adhere to the regimen

SECONDARY OUTCOMES:
Development of AE | 2 years
  Cumulative incidence of AE
Transepidermal water loss | 2 years
  Development of transepidermal water loss over time
Microbiome diversity | 2 years
  Development of microbiome diversity over time

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Weidinger, Prof, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- USchleswig-Holstein, Kiel, Scheswig-Holstein, Germany